CLINICAL TRIAL: NCT05269316
Title: A First-in-human, Phase 1/2, Open-label, Multi-center, Dose-escalation and Dose-expansion Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Anti-tumor Activity of the ATR Inhibitor IMP9064 Monotherapy and in Combination With PARP Inhibitor Senaparib in Patients With Advanced Solid Tumors
Brief Title: Study to Evaluate IMP9064 as a Monotherapy or in Combination in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Impact Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IMP9064-101
Record Dates: First submitted 2022-02-11; First posted 2022-03-07 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-08

CONDITIONS: Solid Tumor; Advanced Solid Tumor
Keywords: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- IMP9064 Monotherapy (Experimental): Dose-escalation IMP9064 administered orally on empty stomach once/twice daily
  Interventions: Drug: IMP9064

INTERVENTIONS:
Drug: IMP9064 — IMP9064 Monotherapy administered for 21 days

SUMMARY:
This is a Phase 1/2, multicenter, open-label study to evaluate the safety and efficacy of IMP9064 as monotherapy or in combination with PARP inhibitor Senaparib in patients with advanced solid tumors

DETAILED DESCRIPTION:
IMP9064 is an investigational therapeutic protein that may prevent repair of DNA damage in tumor cell. IMP9064 acts as inhibitor (blocker)of the proteins ataxia-telangiectasia and Rad3-related kinase (ATR) which are important in cancer cell DNA repair. If cancer cells cannot repair damage to their DNA, then there is a high possibility that cancer cells will not survive.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years of age on the day of signing informed consent form (ICF) (at the time of screening for Part 1 and Part 2C and pre-screening for Part 2A and Part 2B).
2. Must voluntarily participate in the study and be willing and able to provide signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.
3. Male or female patients with histologically or cytologically confirmed AST refractory to or intolerant of available standard-of-care therapy or for which no standard treatment exists.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1 (Part 1) at screening.
5. Provision of tumor tissue samples.
6. Life expectancy ≥ 12 weeks (according to Investigator's judgement).
7. Female patients should meet at least 1 of the following criteria before they can participate in the study:

   1. Females who have no childbearing potential (i.e. physiologically incapable of pregnancy), including those who have undergone hysterectomy, bilateral oophorectomy, or bilateral salpingectomy.
   2. Post-menopausal (total cessation of menses for ≥ 1 year).
   3. Females of childbearing potential should have a negative serum pregnancy test during the screening period (within 7 days prior to the first dose of the study drug), should not be in lactation, and should be willing to practice a highly effective contraceptive method throughout the study period (from study entry up to 6 months after the last dose of the study drug). A highly effective method of contraception is defined as one that results in a low failure rate, i.e., less than 1% per year, when used consistently and correctly (See Appendix 4, Section 11.4).
8. Male patients are eligible to participate in the study if they have undergone vasectomy or agree to use a highly effective method of contraception and refrain from donating sperms from study entry up to 6 months after the last dose of the study drug.
9. Willing and able to comply with study visits and study-related procedures.
10. For optional PD analysis in Part 1, patients should be willing provide hairs plucked from eyebrows pre and post treatment with IMP9064 and fresh tumor biopsies (if deemed necessary by SMC) pre and post treatment with IMP9064.

Exclusion Criteria:

1. Known history of hypersensitivity to any components of the study drug.
2. Any investigational or approved systemic cancer therapy (including chemotherapy, immunotherapy, hormonal therapy and herbal/alternative therapies with anti-cancer indications, or targeted therapy) administered within 28 days or 5 half-lives, whichever is shorter, before the first dose of study drug.
3. Any previous treatment-related toxicities have not recovered, i.e. to ≤ Grade 1, as evaluated by NCI-CTCAE version 5.0 or baseline, except alopecia and anemia. Patients with chronic Grade 2 toxicities which are well managed and stable may be eligible per the discretion of the investigator after the discussion with the Sponsor and medical monitor, e.g., Grade 2 chemotherapy-induced neuropathy.
4. Primary tumor in CNS, or active or untreated CNS metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are clinically stable for at least 28 days and have no evidence of new or enlarging brain metastases and no requirements for high-dose corticosteroids 14 days prior to dosing with study drug. Patients on low dose corticosteroids (< 20 mg prednisone or equivalent per day) may participate.
5. Clinically significant cardiovascular condition, including:

   * History of congestive heart failure (New York Heart Association [NYHA] Class > 2)
   * History of unstable angina
   * New-onset angina or myocardial infarction within the 6 months prior to the first dose of study drug
   * New onset of atrial fibrillation, supraventricular arrhythmia, or ventricular arrhythmia within the 6 months prior to the first dose of study drug and requiring treatment or intervention. History of atrial fibrillation, supraventricular arrhythmia, or ventricular arrhythmia will be allowed provided the condition is stably controlled.
6. History or presence of an abnormal ECG that, in the Investigator's opinion, is clinically meaningful (including QTcF > 470 msec for females, QTcF > 450 msec for males by Fridericia formula at screening, pacemaker installation or previous diagnosis of congenital long QT syndrome).
7. Patients who have undergone a major surgery or have undergone a radical radiotherapy within 28 days prior to the first dose of study drug or have undergone a palliative radiotherapy within 14 days prior to the first dose of study drug, or have used a radioactive drug (Strontium, Samarium, etc.) within 56 days prior to first dose of study drug.
8. Patients with infections, including:

   * An uncontrolled acute infection, or an active infection requiring systemic treatment, or patients who have received systemic antibiotics within 14 days prior to the first dose of the study drug; prophylaxis use of systemic antibiotics treatment for upper tract infection is allowed as long as there is no violation with the requirement of concomitant medications.
   * A known history of human immunodeficiency virus (HIV) infection and/or acquired immunodeficiency syndrome or positive HIV testing should undergo CD4+ T-cell test during the screening period. Patients with CD4+ T-cell counts < 350 cells/μL are ineligible for enrolment as well as patients with unknown HIV infection status who are unwilling to undergo HIV testing.
   * A known active hepatitis B or C. To be included in the study, patients with hepatitis B virus surface antigen (HBsAg) or hepatitis C virus (HCV) antibody positive test results during screening must be further tested for hepatitis B virus (HBV) DNA titer (excluding patients with a DNA titer of more than 2500 copies [cps]/mL or 500 IU/mL) and HCV ribonucleic acid (RNA) (excluding patients with an HCV RNA concentration exceeding the lower detection limit of the assay) to exclude active hepatitis B or hepatitis C infection requiring treatment. Hepatitis B virus carriers, patients with stable hepatitis B infection after drug treatment (DNA titer not exceeding 2500 copies [cps]/mL or 500 IU/mL) and hepatitis C infected patients who received treatment and achieved sustained virologic response for at least 12 weeks can be enrolled. Note: If the lower detection limit of the HBV DNA assay is higher than 2500 copies [cps]/mL or 500 IU/mL, the patients with an HBV DNA assay result lower than the lower detection limit of the assay can be enrolled.
   * Active tuberculosis.
9. Positive test result for severe acute respiratory syndrome-related coronavirus (SARS-CoV-2) test. SARS-CoV-2 test is mandatory during screening for patients who have exposure to suspected, probable, or confirmed cases of SARS-CoV-2 infection within 14 days, via a validated test per local guidance; the result should be available within 4 days prior to the first dose of study drug.
10. Any other medical (e.g., Child-Pugh class B or C, pulmonary, metabolic, congenital, endocrinal or CNS disease, etc.), psychiatric, or social condition deemed by the Investigator to be likely to interfere with a patient's rights, safety, welfare or ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results.
11. Receipt of:

    * Any treatment targeting the ATR/CHK1 pathway.
    * Live virus or bacterial vaccine within 28 days prior to the first dose of study drug and whilst the patient is receiving study drug. Patients who require COVID-19 vaccination whilst on study drug should receive a non-live vaccine (e.g., one based on messenger RNA (mRNA) or fully inactivated/genetically modified viruses incapable of replication) (see Section 6.8.1).
12. Participation in another clinical study with an investigational product administered in the last 28 days or 5 half-lives (whichever is shorter) prior to the first administration of study drug.
13. An investigational device within 28 days prior to the first dose of study drug.
14. Patients who may need continuous treatment with proton pump inhibitors or potassium competitive acid blockers during the study period.
15. Patients who have other malignancies requiring treatment within 2 years prior to the first dose of study drug will be excluded, except for radically treated locally curable basal or squamous cell skin cancer and other malignancies that have been treated with no relapse within 2 years. Presence of other active invasive cancers will be excluded for Part 2.
16. Patients who are unable to swallow oral medications.
17. Patients who have gastrointestinal illnesses that may affect the absorption of oral medications.
18. Patients with a previously documented diagnosis of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML), or patients who have received transplantation including patients with previous allogeneic bone marrow transplant.
19. Patients known to have a history of alcoholism or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2022-02-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (Safety and Tolerability) | 11 months
  Safety and tolerability as determined by the incidence of adverse events (AEs), including severe AEs and serious AEs (SAEs)
To determine the Maximum Tolerable Dose | 11 months
  Maximum Tolerable Dose (if any)/Recommended Phase 2 Dose of IMP9064 monotherapy

SECONDARY OUTCOMES:
To determine Maximum concentration (Cmax) | 11 months
  The plasma concentration data of IMP9064 from this study will be analyzed using a non-linear mixed effects modeling (NONMEM)
To determine area under the concentration-time curve from time zero to the time of the last quantifiable concentration (AUC0-t) | 11 months
  The plasma concentration data of IMP9064 from this study will be analyzed using a non-linear mixed effects modeling (NONMEM)
To assess Overall response rate (ORR) | 11 months
  Anti-tumor activity of IMP9064 monotherapy assessed as Overall response rate (ORR) according to RECIST version 1.1 in AST patients
To assess Disease control rate (DCR) | 11 months
  Anti-tumor activity of IMP9064 monotherapy assessed as Disease control rate (DCR) according to RECIST version 1.1 in AST patients
To assess Duration of response(DOR) | 11 months
  Anti-tumor activity of IMP9064 monotherapy assessed as Duration of response(DOR) according to RECIST version 1.1 in AST patients
To assess Progression free survival(PFS) | 11 months
  Anti-tumor activity of IMP9064 monotherapy assessed as Progression free survival(PFS) according to RECIST version 1.1 in AST patients
To assess Overall survival(OS) | 11 months
  Anti-tumor activity of IMP9064 monotherapy assessed as Overall survival(OS) according to RECIST version 1.1 in AST patients
To assess QT interval | 11 months
  To assess correlation between plasma concentrations of IMP9064 and QT interval

CONTACTS AND LOCATIONS:
Locations (8):
- United States (4):
  - Hackensack University Medical Center PARTNER, Hackensack, New Jersey
  - Mount Sinai, New York, New York
  - Greenville Hospital System University Medical Center (ITOR), Greenville, South Carolina
  - Mary Crowley Cancer Research Centers, Dallas, Texas
- Australia (2):
  - Blacktown Hospital, Blacktown, New South Wales
  - Linear Clinical Research Limited, Nedlands
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No